CLINICAL TRIAL: NCT00219479
Title: Dilantin Levels With Continuous Delivery of Enteral Feedings - A Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting subjects
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #96-264
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Seizures
Keywords: seizure prophylaxis; enteral nutrition
MeSH Terms: conditions — Seizures | interventions — Phenytoin; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Phenytoin (Dilantin) levels during change in enteral feeding

SUMMARY:
It is unclear how enteral nutrition via a feeding tube should be given when a patient is receiving enteral Dilantin. Some caregivers hold the feedings for one hour before and one hour after the Dilantin dose to insure adequate absorption of the medication and some caregivers think that the feedings do not need to be interrupted.

Hypothesis: Dilantin levels will remain therapeutic when enteral nutrition is given continuously during the administration of enteral Dilantin.

The objective of this study is to determine Dilantin levels when enteral feedings are given by the continuous method. Thirty patients will be studied. When Dilantin levels are in the therapeutic range for 2 consecutive days on interrupted feedings (baseline), the patient will be switched to continuous feedings uninterrupted for the medication, for 7 days. Dilantin levels will be checked daily and if the levels become subtherapeutic an intravenous (IV) bolus of Dilantin will be given and the enteral dose will be increased (doses determined by primary caregiver). Serum albumin will be measured at baseline and at the beginning and end of each week, in order to calculate free Dilantin.

DETAILED DESCRIPTION:
Rationale: It is unclear how enteral nutrition via feeding tube should be given when a patient is receiving enteral Dilantin. Some caregivers hold the feedings for one hour before and one hour after the Dilantin dose to insure adequate absorption of the medication and some caregivers think that the feedings do not need to be interrupted. Both methods are used in this institution, although the interrupted method is recommended by the Clinical Nutrition Service. Interrupting the feedings has the obvious disadvantage that the patient receives less hours of feeding and requires more nursing intervention.

Key Objectives: To determine the change in Dilantin levels when enteral feedings are given by the continuous method.

Study Population: 30 patients already on Dilantin for seizure prophylaxis who are already receiving enteral nutrition by the interrupted method and have stable, therapeutic Dilantin levels.

Major Inclusion Criteria:

1. on Dilantin for seizure prophylaxis (dose determined by primary caregiver) with therapeutic Dilantin levels
2. receiving enteral nutrition by the interrupted method at goal feeding rate;
3. age >18
4. feeding tube in proper position, no restriction as to type of feeding tube (nasogastric, nasoduodenal, gastrostomy, jejunostomy), but both Dilantin and enteral feeding must be given through the same tube.

Major Exclusion Criteria:

1. history of seizures
2. albumin infusions necessary during study period
3. anticipation that feedings will need to be held for more than 4 hours at a time
4. Patients that do not maintain stable Dilantin levels (< 25% variability) with the interrupted method of feeding; 5) inability to obtain consent from patient or spokesperson.

Allocation to Groups: all patients will be switched from baseline method of feeding (interrupted) to continuous feeding.

Procedures: When Dilantin levels are in the therapeutic range for 2 consecutive days on interrupted feedings (baseline), the patient will be switched to continuous feedings uninterrupted for the medication, for 7 days. Dilantin levels will be checked daily and if the levels become subtherapeutic an IV bolus of Dilantin will be given and the enteral dose will be increased (doses determined by primary caregiver). Serum albumin will be measured at baseline and at the beginning and end of each week, in order to calculate free Dilantin.

Risks and Discomforts:

1. subtherapeutic Dilantin levels, but these will be closely followed;
2. seizures, patient will be discontinued if this occurs;
3. venipuncture for 10 Dilantin levels and 3 serum albumin determinations (minimum blood for each test is 0.4 cc).

Confidentiality: Subjects will be identified only by initials and study number.

ELIGIBILITY:
Inclusion Criteria:

1. On Dilantin for seizure prophylaxis (dose determined by primary caregiver) with therapeutic Dilantin levels
2. Receiving enteral nutrition by the interrupted method at goal feeding rate
3. Age >18
4. Feeding tube in proper position, no restriction as to type of feeding tube (nasogastric, nasoduodenal, gastrostomy, jejunostomy), but both Dilantin and enteral feeding must be given through the same tube

Exclusion Criteria:

1. History of seizures
2. Albumin infusions necessary during study period
3. Anticipation that feedings will need to be held for more than 4 hours at a time
4. Patients that do not maintain stable Dilantin levels (< 25% variability) with the interrupted method of feeding
5. Inability to obtain consent from patient or spokesperson

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1997-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Dilantin levels

CONTACTS AND LOCATIONS:
Overall Officials: Sandralee A Blosser, MD, Principal Investigator — Penn State University